CLINICAL TRIAL: NCT04293055
Title: Examination of Phone Coaching as a Weight Loss Maintenance Strategy
Brief Title: Phone Coaching for Weight Loss Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Jessica Unick, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1561299
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Weight Loss
Keywords: Phone coaching; Diet; Exercise
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance program+possibility of phone coaching (Experimental): All participants are provided with a monthly newsletter which contains useful strategies for maintaining weight loss long-term. Participants are also encouraged to weigh themselves daily using a smart scale, which electronically transmits weight data to the research staff. Some participants randomized to this condition will also receive 4 consecutive weeks of phone coaching at some point over the 1-year intervention period (this is determined by a weight-based algorithm).
  Interventions: Behavioral: Maintenance program; Behavioral: Phone coaching
- Maintenance program only (Active Comparator): All participants are provided with a monthly newsletter which contains useful strategies for maintaining weight loss long-term. Participants are also encouraged to weigh themselves daily using a smart scale, which electronically transmits weight data to the research staff. No participants in this condition will receive phone coaching.
  Interventions: Behavioral: Maintenance program

INTERVENTIONS:
Behavioral: Maintenance program — 1-year weight loss maintenance program, consisting of monthly newsletters
Behavioral: Phone coaching — Some individuals will receive 4 consecutive weeks of phone coaching. The first coaching call will be approximately 30 minutes in duration and follow-up calls will be 10-15 minutes in duration. Coaches will help support participants in their weight loss maintenance efforts. Once coaching calls are completed, the participant will not have any other contact with their coach.
  Arms: Maintenance program+possibility of phone coaching

SUMMARY:
The purpose of this study was to examine whether 4 consecutive weeks of phone coaching aids in recovery from weight regain during weight loss maintenance. Individuals who previously achieved and maintained a >=5% weight loss in a 1-year behavioral weight loss program were provided with a low-intensity maintenance intervention (monthly newsletters and smart scale). At baseline, participants were randomized to the coaching group or the control group (no coaching). If participants regained >1.5% of their weight, randomization was "triggered." At this point, participants randomized to the coaching condition received 4 brief weekly coaching calls; participants randomized to the control condition received no additional intervention contact. Short-term and long-term weight change was assessed and compared between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* 18-72 years of age
* Recent completion of a 1-year behavioral weight loss program
* Achievement of >=5% weight loss at the end of the 1-year weight loss program

Exclusion Criteria:

* Not currently enrolled in another weight management program

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Unick, PhD, Principal Investigator — The Miriam Hospital's Weight Control and Diabetes Research Center
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hayes JF, Ross KM, Pellegrini C, Wing RR, Webster J, Derrick A, Tobin SY, Unick JL. Brief coaching intervention to reverse weight regain during weight loss maintenance: a preliminary randomized controlled trial. J Behav Med. 2025 Aug;48(4):706-714. doi: 10.1007/s10865-025-00582-x. Epub 2025 Jun 26. PMID 40569564

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Maintenance Program+Possibility of Phone Coaching | Maintenance Program Only
Started | 41 | 36
Triggered Randomization | 35 | 31
Received Randomization Condition | 33 (Study ended prior to full coaching dose (n=2)) | 31
Completed | 34 | 30
Not Completed | 7 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Did not trigger randomization | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maintenance Program+Possibility of Phone Coaching | Maintenance Program Only | Total
Number analyzed (Participants) | 41 | 36 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (10.5) | 56.4 (8.7) | 54.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 38 | 33 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 3 | 3 | 6
  White | 34 | 30 | 64
  Other | 2 | 0 | 2
  More than One Race | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 41 | 36 | 77
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (4.4) | 29.1 (3.9) | 29.2 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Body Weight From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: Only individuals who regained 1.5% weight and triggered randomization condition were included in the analysis. Multiple imputation used to correct for missing data.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Maintenance Program+Possibility of Phone Coaching | Maintenance Program Only
Number analyzed (Participants) | 35 | 31
percent change | 5.18 (0.72) | 5.71 (0.76)

2. Secondary Outcome: Percent Weight Change Over the Coaching Period
Description: The 'coaching period' weight change was calculated by subtracting the 'trigger date' weight (i.e., the weight measurement from the smart scale on the day the participant achieved the trigger threshold, which was defined as the final day in a series of 4 days >1.5% or the final day in which the previous 7 days averaged >1.5%) from the smart scale weight 40 days following the 'trigger date'. Percent weight change was then calculated by taking the 'coaching period weight change' and dividing it by the 'trigger date weight' and multiplying by 100. Therefore, a negative number indicates weight loss and a positive number indicates weight gain over the 40-day coaching period.
Time Frame: Trigger date and 40 days post-trigger date
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Maintenance Program+Possibility of Phone Coaching | Maintenance Program Only
Number analyzed (Participants) | 35 | 31
percent change | -1.05 (0.3) | 0.37 (0.31)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Maintenance Program+Possibility of Phone Coaching | Maintenance Program Only
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/36
Other Adverse Events (participants affected / at risk) | 0/41 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT04293055/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT04293055/SAP_001.pdf